CLINICAL TRIAL: NCT00844805
Title: Infliximab as First Line Therapy in Patients With Early Active Axial Spondyloarthritis Trial
Brief Title: Infliximab for Treatment of Axial Spondyloarthritis (P05336 AM1)
Acronym: INFAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05336; 2008-000982-51
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Ankylosing Spondylitis; Axial Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — Infliximab; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Infliximab + Naproxen (Experimental): Infliximab administered at a dose of 5 mg/kg intravenously on Day 1 of Weeks 0, 2, 6, 12, 18, and 24, combined with naproxen administered at a daily dose of 1000 mg for 28 weeks during the 28-week treatment phase.
  Interventions: Drug: Infliximab; Drug: Naproxen
- Placebo + Naproxen (Placebo Comparator): Placebo administered intravenously on Day 1 at Weeks 0, 2, 6, 12, 18, and 24, combined with naproxen administered at a daily dose of 1000 mg for 28 weeks, during the 28-week treatment phase.
  Interventions: Drug: Placebo; Drug: Naproxen
- Naproxen Only (Follow-Up) (Experimental): For participants who achieved partial remission during 28-week treatment phase, naproxen was continued at a daily dose of 1000 mg administered orally for an additional 24 weeks in the follow-up phase.
  Interventions: Drug: Naproxen
- No Treatment (Follow-Up) (No Intervention): For participants who achieved partial remission during Treatment phase, no treatment was administered for an additional 24 weeks in the follow-up phase.

INTERVENTIONS:
Drug: Infliximab
  Other Names: Remicade; SCH 215596
  Arms: Infliximab + Naproxen
Drug: Placebo
  Arms: Placebo + Naproxen
Drug: Naproxen
  Other Names: Naprosyn
  Arms: Infliximab + Naproxen; Naproxen Only (Follow-Up); Placebo + Naproxen

SUMMARY:
The primary objective of this study was to assess the proportion of participants in the infliximab plus naproxen arm versus the placebo plus naproxen arm, in a population of participants with moderate-to-severe active axial spondyloarthritis and disease duration of ≤3 years, who achieve the Assessment in Ankylosing Spondylitis (ASAS) partial remission criteria.

DETAILED DESCRIPTION:
In the 28-week treatment phase, participants were randomized to receive either infliximab plus naproxen or placebo plus naproxen.

After 28-weeks of treatment, participants that achieved partial remission in the treatment phase were randomized to continued treatment with naproxen or to receive no treatment and were followed for an additional 24 weeks (follow-up phase).

ELIGIBILITY:
Inclusion Criteria:

Participant must:

* be 18 to 48 years of age
* have diagnosis of active axial spondyloarthritis, with disease duration of less than or equal to 3 years.
* have active disease during trial enrollment
* have limited treatment history for axial spondyloarthritis (must meet certain criteria)
* agree to an acceptable method of contraception (for women of childbearing potential and all men)
* must meet certain tuberculosis screening requirements
* must meet certain laboratory screening safety requirements
* have an x-ray of the sacroiliac joints available from within the previous 12 months (or have one performed during the Screening visit if site is outside of Germany).

Exclusion Criteria:

Participant will be excluded:

* for certain medical conditions and/or recent history of certain medical disorders
* for current or recent treatment with certain other medications and certain vaccinations.
* for being a woman who is breastfeeding, pregnant, or intending to become pregnant.
* if known to have had a substance abuse problem within the previous 3 years prior to screening.
* if currently participating in any other clinical study.
* for other administrative reasons.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sieper J, Lenaerts J, Wollenhaupt J, Rudwaleit M, Mazurov VI, Myasoutova L, Park S, Song Y, Yao R, Chitkara D, Vastesaeger N; All INFAST Investigators. Efficacy and safety of infliximab plus naproxen versus naproxen alone in patients with early, active axial spondyloarthritis: results from the double-blind, placebo-controlled INFAST study, Part 1. Ann Rheum Dis. 2014 Jan;73(1):101-7. doi: 10.1136/annrheumdis-2012-203201. Epub 2013 May 21. PMID 23696633
- [Result] Sieper J, Lenaerts J, Wollenhaupt J, Rudwaleit M, Mazurov VI, Myasoutova L, Park S, Song Y, Yao R, Chitkara D, Vastesaeger N; All INFAST Investigators. Maintenance of biologic-free remission with naproxen or no treatment in patients with early, active axial spondyloarthritis: results from a 6-month, randomised, open-label follow-up study, INFAST Part 2. Ann Rheum Dis. 2014 Jan;73(1):108-13. doi: 10.1136/annrheumdis-2013-203460. Epub 2013 Jun 5. PMID 23740231
- [Derived] Poddubnyy D, Listing J, Sieper J. Brief Report: Course of Active Inflammatory and Fatty Lesions in Patients With Early Axial Spondyloarthritis Treated With Infliximab Plus Naproxen as Compared to Naproxen Alone: Results From the Infliximab As First Line Therapy in Patients with Early Active Axial Spondyloarthritis Trial. Arthritis Rheumatol. 2016 Aug;68(8):1899-903. doi: 10.1002/art.39690. PMID 27015283

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Naproxen: Placebo administered intravenously on Day 1 of Weeks 0, 2, 6, 12, 18, and 24, combined with naproxen administered at a daily dose of 1000 mg for 28 weeks, during the 28-week treatment phase.
- Naproxen: For participants who achieved partial remission during 28-week treatment phase, naproxen was continued at a daily dose of 1000 mg administered orally for an additional 24 weeks in the follow-up phase.
- No Treatment: For participants who achieved partial remission during Treatment phase, no treatment was administered for an additional 24 weeks in the follow-up phase.
Period: Treatment Phase
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen | Naproxen | No Treatment
Started | 106 | 52 | 0 | 0
Completed | 96 | 45 | 0 | 0
Not Completed | 10 | 7 | 0 | 0
Not completed — Adverse Event | 5 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 0 | 0
Not completed — Noncompliance With Protocol | 1 | 0 | 0 | 0
Not completed — Did Not Meet Protocol Eligibility | 1 | 2 | 0 | 0
Period: Follow-Up Phase
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen | Naproxen | No Treatment
Started | 0 | 0 | 41 (Participants who met partial remission criteria at the end of treatment entered the Follow-Up Phase.) | 41 (Participants who met partial remission criteria at the end of treatment entered the Follow-Up Phase.)
Completed | 0 | 0 | 32 | 32
Not Completed | 0 | 0 | 9 | 9
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 3
Not completed — Noncompliance With Protocol | 0 | 0 | 0 | 1
Not completed — Relapse/Recurrence | 0 | 0 | 2 | 4
Not completed — Did Not Meet Protocol Eligibility | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen | Total
Number analyzed (Participants) | 105 | 51 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age presented is based on the Intent-to-Treat (ITT) population which consisted of participants treated with Infliximab + Naproxen (n=105) and participants treated with Placebo + Naproxen (n=51).
  years | 31.7 (8.51) | 30.7 (7.34) | 31.4 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender is based on the Intent-to-Treat (ITT) population which consisted of participants treated with Infliximab + Naproxen (n=105) and participants treated with Placebo + Naproxen (n=51).
  Participants
    Female | 33 | 11 | 44
    Male | 72 | 40 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving the Assessment in Ankylosing Spondylitis (ASAS) Partial Remission Criteria at Week 28
Description: ASAS domains were measured on a visual analog scale (VAS) of 0 to 100 mm (with 0 being the very best situation and 100 being the very worst situation). ASAS partial remission criteria is defined as reaching ≤20 mm in all 4 ASAS domains (i.e., patient global assessment, total back pain, function, and inflammation).
Time Frame: Week 28
Population: The Intent-to-Treat Population consisted of all participants who were randomized, took at least one dose of study medication, and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 105 | 51
Participants
  Achieved Partial Remission | 65 | 18
  Did Not Achieve Partial Remission | 40 | 33

2. Secondary Outcome: Number of Participants Maintaining the ASAS Partial Remission Criteria at Week 52 By Treatment Assignment in the Follow-Up Phase
Description: ASAS domains were measured on a VAS of 0 to 100 mm (with 0 being the very best situation and 100 being the very worst situation). ASAS partial remission criteria is defined as reaching ≤20 mm in all 4 ASAS domains (i.e., patient global assessment, total back pain, function, and inflammation).
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Naproxen: For participants who achieved remission during 28-week treatment phase, naproxen was continued at a daily dose of 1000 mg administered orally for an additional 24 weeks in the follow-up phase.
- No Treatment: For participants who achieved remission during Treatment phase, no treatment was administered for an additional 24 weeks in the follow-up phase.
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 40 | 40
Participants
  Achieved Partial Remission | 19 | 16
  Did Not Achieve Partial Remission | 21 | 24

3. Secondary Outcome: Percentage of Participants Maintaining the ASAS Partial Remission Criteria at Week 52 By Treatment Assignment in the Treatment Phase
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 105 | 51
Percentage of Participants | 40 | 55

4. Secondary Outcome: Change From Baseline of Berlin Magnetic Resonance Imaging (MRI) Spine Overall Score at Week 28
Description: MRI scans (T1 for chronic changes and short tau inversion recovery [STIR] for active changes) of the whole spine was performed to determine the Berlin MRI Spine Score. The Berlin MRI scoring for the spine was assessed on a scale of 0 (best) to 3 (worst) for a maximum total score of 69, with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable.
Time Frame: Baseline, Week 28
Population: The number of participants represented those with a screening value and a value at treatment Week 28.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 98 | 47
Units on a Scale | -0.5 [-3.5 to 0.0] | 0.0 [-4.7 to 0.0]

5. Secondary Outcome: Change From Baseline in the Sacroiliac Overall Score at Week 28
Description: Each sacroiliac joint was divided into four quadrants. An activity score of 0 (best) to 3 (worst) was assessed for every quadrant of the left and right sacroiliac joint separately for a total maximum score of 24, with with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable.
Time Frame: Baseline, Week 28
Population: The number of participants represented those with a screening value and a value at treatment Week 28.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 97 | 47
Units on a Scale | -2.0 [-7.0 to -0.5] | -3.0 [-6.5 to -1.0]

6. Secondary Outcome: Change From Baseline of Berlin MRI Spine Overall Score at Week 52
Description: MRI scans (T1 for chronic changes and STIR for active changes) of the whole spine was performed to determine the Berlin MRI Spine Score. The Berlin MRI scoring for the spine was assessed on a scale of 0 (best) to 3 (worst) for a maximum total score of 69, with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable.
Time Frame: Baseline, Week 52
Population: The number of participants represents those with a Week 28 values and those with a Week 52 value.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 37 | 37
Units on a Scale | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 2.3]

7. Secondary Outcome: Change From Baseline in the Sacroiliac Overall Score at Week 52
Description: as for outcome 5
Time Frame: Baseline, Week 28
Population: The number of participants represented those with a screening value and a value at treatment Week 28.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 36 | 36
Units on a Scale | 1.1 [0.0 to 4.0] | 1.0 [0.0 to 3.3]

8. Secondary Outcome: Number of Participants With Complete Absence of Active Inflammatory Lesions at the Spine at Treatment Week 28
Description: MRI scans (T1 for chronic changes and STIR for active changes) of the whole spine was performed to determine the Berlin MRI Spine Score. The Berlin MRI scoring for the spine was assessed on a scale of 0 (best) to 3 (worst) for a maximum total score of 69, with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable. Complete absence of active inflammatory lesions was defined as a Berlin MRI Score = 0.
Time Frame: Week 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 105 | 51
Participants | 63 | 23
Statistical Analysis 1: Comparison: Infliximab + Naproxen vs Placebo + Naproxen; Test type: Superiority or Other; p = 0.0884, Fisher Exact; Difference in Percentages = 14.9, 95% CI 2-sided [-1.7 to 31.5] — The 95% CI for treatment differences were computed using Wilson's Method

9. Secondary Outcome: Number of Participants With Complete Absence of Active Inflammatory Lesions at the Sacroiliac Joint at Treatment Week 28
Description: Each sacroiliac joint was divided into four quadrants. An activity score of 0 (best) to 3 (worst) was assessed for every quadrant of the left and right sacroiliac joint separately for a total maximum score of 24, with with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable. Complete absence of active inflammatory lesions at the sacroiliac joints was defined as a Score = 0.
Time Frame: Week 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 105 | 51
Participants | 29 | 3
Statistical Analysis 1: Comparison: Infliximab + Naproxen vs Placebo + Naproxen; Test type: Superiority or Other; p = 0.0013, Fisher Exact; Difference in Percentages = 21.7, 95% CI 2-sided [11.0 to 32.5] — The 95% CI for treatment differences were computed using Wilson's Method

10. Secondary Outcome: Number of Participants With Complete Absence of Active Inflammatory Lesions at the Spine and Sacroiliac Joint at Treatment Week 28
Description: MRI scans (T1 for chronic changes and STIR for active changes) of the whole spine was performed to determine the Berlin MRI Spine Score. The Berlin MRI scoring for the spine was assessed on a scale of 0 (best) to 3 (worst) for a maximum total score of 69, with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable. Complete absence of active inflammatory lesions was defined as a Berlin MRI Score = 0.
  Each sacroiliac joint was divided into four quadrants. An activity score of 0 (best) to 3 (worst) was assessed for every quadrant of the left and right sacroiliac joint separately for a total maximum score of 24, with with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable. Complete absence of active sacroiliac inflammatory lesions was defined as a Score = 0.
Time Frame: Week 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 105 | 51
Participants | 19 | 0
Statistical Analysis 1: Comparison: Infliximab + Naproxen vs Placebo + Naproxen; Test type: Superiority or Other; p = 0.0004, Fisher Exact; Difference in Percentages = 18.1, 95% CI 2-sided [10.7 to 25.5] — The 95% CI for treatment differences were computed using Wilson's Method

11. Secondary Outcome: Number of Participants With Complete Absence of Active Inflammatory Lesions at the Spine at Treatment Week 52
Description: as for outcome 8
Time Frame: Week 52
Population: The Intent-to-Treat Population consisted of all participants that were randomized, took at least one dose of study medication, and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 40 | 40
Participants | 20 | 16
Statistical Analysis 1: Comparison: Naproxen vs No Treatment; Test type: Superiority or Other; p = 0.5005, Fisher Exact; Difference in Percentages = 10.0, 95% CI 2-sided [-11.7 to 31.7] — The 95% CI for treatment differences were computed using Wilson's Method

12. Secondary Outcome: Number of Participants With Complete Absence of Active Inflammatory Lesions at the Sacroiliac Joint at Treatment Week 52
Description: EaEach sacroiliac joint was divided into four quadrants. An activity score of 0 (best) to 3 (worst) was assessed for every quadrant of the left and right sacroiliac joint separately for a total maximum score of 24, with with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable. Complete absence of active sacroiliac inflammatory lesions was defined as a Score = 0.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 40 | 40
Participants | 3 | 4
Statistical Analysis 1: Comparison: Naproxen vs No Treatment; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Difference in Percentages = -2.5, 95% CI 2-sided [-14.9 to 9.9] — The 95% CI for treatment differences were computed using Wilson's Method

13. Secondary Outcome: Number of Participants With Complete Absence of Active Inflammatory Lesions at the Spine and Sacroiliac Joint at Treatment Week 52
Description: MRI scans (T1 for chronic changes and STIR for active changes) of the whole spine was performed to determine the Berlin MRI Spine Score. The Berlin MRI scoring for the spine was assessed on a scale of 0 (best) to 3 (worst) for a maximum total score of 69, with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable. Complete absence of active spinal inflammatory lesions was defined as a Berlin MRI Score = 0.
  Each sacroiliac joint was divided into four quadrants. An activity score of 0 (best) to 3 (worst) was assessed for every quadrant of the left and right sacroiliac joint separately for a total maximum score of 24, with with 0 = no inflammatory lesions; 1 = minor bone marrow edema; 2 = moderate bone marrow edema; 3 = major bone marrow edema; or N = non readable. Complete absence of active sacroiliac inflammatory lesions was defined as a Score = 0.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 40 | 40
Participants | 1 | 1
Statistical Analysis 1: Comparison: Naproxen vs No Treatment; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Difference in Percentages = 0.0, 95% CI 2-sided [-6.8 to 6.8] — The 95% CI for treatment differences were computed using Wilson's Method

14. Secondary Outcome: Median Duration of Maintaining ASAS Partial Remission in the Follow-Up Phase
Description: ASAS domains were measured on a VAS of 0 to 100 mm (with 0 being the very best situation and 100 being the very worse situation). ASAS partial remission criteria is defined as reaching ≤20 mm in all 4 ASAS domains (i.e., patient global assessment, total back pain, function, and inflammation).
Time Frame: Week 52
Population: The Intent-to-Treat Population consisted of all participants who were randomized to treatment, took at least one dose of study medication, and had at least one post-baseline efficacy assessment.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 40 | 40
Weeks | 23.00 [3.43 to 26.71] | 12.57 [4.71 to 25.14]
Statistical Analysis 1: Comparison: Naproxen vs No Treatment; Test type: Superiority or Other; p = 0.3802, Log Rank

15. Secondary Outcome: Number of Participants Who Achieved ASAS Partial Remission That Experienced Disease Flare With Naproxen Maintenance Treatment in the Follow-Up Phase
Description: The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) employs a VAS of 0mm (best) to 100mm (worst). Disease flare was defined as reaching a BASDAI of ≥30 mm during two consecutive visits after Week 28 until Week 52.
  ASAS domains were measured on a VAS of 0 to 100 mm (with 0 being the very best situation and 100 being the very worse situation). ASAS partial remission criteria was defined as reaching ≤20 mm in all 4 ASAS domains (i.e., patient global assessment, total back pain, function, and inflammation).
Time Frame: Week 52
Population: The Intent-to-Treat Population consisted of all subjects who were randomized, took at least one dose of study medication, and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Naproxen | No Treatment
Number analyzed (Participants) | 40 | 40
Participants | 1 | 3
Statistical Analysis 1: Comparison: Naproxen vs No Treatment; Test type: Superiority or Other; p = 0.6153, Fisher Exact; Difference in Percentages = -5.0, 95% CI 2-sided [-14.5 to 4.5] — The 95% CI for treatment differences were computed using Wilson's Method

16. Secondary Outcome: Percentage of Participants That Achieved ASAS-40 Response at Week 28 in the Treatment Phase
Description: ASAS domains were measured on a VAS of 0 to 100 mm (with 0 being the very best situation and 100 being the very worse situation). ASAS-40 response was defined as ASAS achieving ≥40% improvement in 3 of the 4 domains (patient global assessment, total back pain, function, and inflammation), with an absolute improvement of ≥20 mm and no deterioration in the remaining domain.
Time Frame: Week 28
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 105 | 51
Percentage of Participants | 79 | 29
Statistical Analysis 1: Comparison: Infliximab + Naproxen vs Placebo + Naproxen; Test type: Superiority or Other; p = 0.0263, Fisher Exact; Difference in Percentages = 18.4, 95% CI 2-sided [2.5 to 34.3] — The 95% CI for treatment differences were computed using Wilson's Method

17. Secondary Outcome: Percentage of Participants That Achieved ASAS-20 Response at Week 28 in the Treatment Phase
Description: ASAS-20 response was defined as ≥20% improvement in response according to following criteria:
  • An improvement of ≥20% from baseline and an absolute improvement from
  baseline of ≥10 mm in at least 3 of the following 4 domains (patient global assessment, pain, function,and inflammation)
  • Absence of deterioration from baseline (≥20% and an absolute change of
  ≥10 mm) in the potential remaining domain.
Time Frame: Week 28
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen
Number analyzed (Participants) | 105 | 51
Percentage of Participants | 85 | 37
Statistical Analysis 1: Comparison: Infliximab + Naproxen vs Placebo + Naproxen; Test type: Superiority or Other; p = 0.3011, Fisher Exact; Difference in Percentages = 8.4, 95% CI 2-sided [-6.0 to 22.8] — The 95% CI for treatment differences were computed using Wilson's Method

ADVERSE EVENTS:
Time Frame: Up to Week 52.
Description: The Safety Population consisted of all participants who received at least one dose of study medication.
Arm/Group | Infliximab + Naproxen | Placebo + Naproxen | Naproxen | No Treatment
Serious Adverse Events (participants affected / at risk) | 6/105 | 3/52 | 0/41 | 3/41
Other Adverse Events (participants affected / at risk) | 24/105 | 8/52 | 6/41 | 11/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Infliximab + Naproxen (N=105) | Placebo + Naproxen (N=52) | Naproxen (N=41) | No Treatment (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carcinoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0/0 (0) | 0 (0) | 0 (0)
Foetal Distress Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine Hypotonus (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab + Naproxen (N=105) | Placebo + Naproxen (N=52) | Naproxen (N=41) | No Treatment (N=41)
Abdominal Pain Upper (Gastrointestinal disorders) | 8 (10) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (7) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (3)
Nasopharyngitis (Infections and infestations) | 13 (16) | 5 (5) | 4 (4) | 6 (9)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 7 (14) | 2 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media. The sponsor shall have the right to review and comment with respect to data analysis and presentation with regard to protected proprietary information, data accuracy, and fair balance.